CLINICAL TRIAL: NCT05290441
Title: Evaluation of Postmortem Pulmonary Interstitial Fibrosis Severity and EGFR Positivity in Covid-19 Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Seyhan Dülger,MD, associate professor, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-KAEK-25 2021/08-10
Record Dates: First submitted 2022-01-13; First posted 2022-03-22 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2022-03

CONDITIONS: Pneumonia, Viral; COVID-19 Pneumonia; EGFR Amplification
MeSH Terms: conditions — Pneumonia, Viral

STUDY DESIGN:
Intervention Model Description: cross-sectional interventional clinical research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- None involement (Active Comparator): In the pathological examination, the group of patients without EGFR involvement in the biopsy material.
  Interventions: Procedure: None involvement
- Mild (Active Comparator): In the pathological examination, the group of patients mild EGFR involvement in the biopsy material.
  Interventions: Procedure: None involvement
- Moderate (Active Comparator): In the pathological examination, the group of patients moderate EGFR involvement in the biopsy material.
  Interventions: Procedure: None involvement
- Severe (Active Comparator): In the pathological examination, the group of patients severe EGFR involvement in the biopsy material
  Interventions: Procedure: None involvement

INTERVENTIONS:
Procedure: None involvement — No EGFR involvement

SUMMARY:
The aim of this study is to examine the relationship between the severity of fibrosis in the lung tissue and EGFR positivity in patients who died due to covid-19 pneumonia, with the demographic characteristics, comorbidities, biochemistry values, treatments they received, and radiological appearances. Transthoracic tru-cut biopsy will be performed on patients who have died in the intensive care unit with the diagnosis of Covid 19 pneumonia. EGFR positivity will be evaluated in the material taken. The relationship between the severity of fibrosis and the demographic data of the patients, the drugs used and their radiological appearances will be analyzed statistically.

DETAILED DESCRIPTION:
The pathophysiology of Covid 19 infection still remains complex. Diffuse alveolo-interstitial damage, organizing pneumonia and severe fibrotic organizing pneumonia have been reported and possibly associated with cytokine storm. However, profibrotic pathways and mediators involved in fibrosis and the severity of fibrosis may differ individually. Epidermal growth factor (EGF) is a protein-structured growth factor that stimulates cell division, differentiation, survival, proliferation, growth and cell migration. It acts through the epidermal growth factor receptor (EGFR). The stimulating effect of fibroblasts, kerotinocytes, and vascular endothelial cells is known to stimulate growth and proliferation, and plays a role in the repair process of the lungs and the development of pulmonary fibrosis. EGFR is also a tyrosine kinase receptor. The relationship between fibrosis severity and EGFR positivity in the tissues of deceased covid pneumonia patients, demographic data of the patients, their combinations and the treatment they receive may guide treatment approaches.

The aim of this study is to examine the relationship between the severity of fibrosis in the lung tissue and EGFR positivity in patients who died due to covid-19 pneumonia, demographic characteristics, comorbidities, biochemistry values, and treatments they receive.

Material methods: Transthoracic tru-cut biopsy will be performed with the permission of their families, for patients hospitalized in the intensive care unit of our hospital and who died due to Covid 19 pneumonia. Biopsy, where the involvement is more intense compared hemithorax to the radiological appearance, will be performed blindly. By studying EGFR on biopsy materials, fibrosis grade will be classified as 0=none; 1=mild; 2=medium; 3=severe. Thoracic CT images of the patients were reviewed by a radiologist, and the fibrosis image and extent will again be classified as 0=none; 1=mild; 2=medium; 3=severe. Medications used, additional diseases, demographic data, length of stay in the intensive care unit, and intubation times will be recorded. The relationship between EGFR positivity and other data will be analyzed statistically.

The relationship between fibrosis severity and EGFR positivity in the tissues of deceased covid pneumonia patients, demographic data of the patients, their combinations and the treatment they receive may guide treatment approaches. It may shed light on the fact that fibrolytic drugs, which act as tyrosine kinase inhibitors and are used in idiopathic interstitial fibrosis, can also be used in covid 19 pneumonia damage.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Patients who died while lying in the Intensive Care Unit with the diagnosis of Covid-19 pneumonia

Exclusion Criteria:

* <18 years old
* Patients who were treated with the diagnosis of Covid 19 pneumonia and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Fibrosis | "through study completion, an average of 1 year".
  EGFR involvement

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Bursa Yüksek İhtisas EAH, Bursa, Eyalet/Yerleşke
  - Seyhan Dülger, Bursa, Yıldırım

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu X, Wang P, Zhang C, Ma Z. Epidermal growth factor receptor (EGFR): A rising star in the era of precision medicine of lung cancer. Oncotarget. 2017 Jul 25;8(30):50209-50220. doi: 10.18632/oncotarget.16854. PMID 28430586
- [Background] George PM, Wells AU, Jenkins RG. Pulmonary fibrosis and COVID-19: the potential role for antifibrotic therapy. Lancet Respir Med. 2020 Aug;8(8):807-815. doi: 10.1016/S2213-2600(20)30225-3. Epub 2020 May 15. PMID 32422178
- [Derived] Dulger SU, Mutlu N, Ceylan I, Ozhan E. The relationship between lung fibrosis, the epidermal growth factor receptor, and disease outcomes in COVID-19 pneumonia: a postmortem evaluation. Clin Exp Med. 2023 Aug;23(4):1181-1188. doi: 10.1007/s10238-022-00872-7. Epub 2022 Aug 20. PMID 35986823